CLINICAL TRIAL: NCT04492397
Title: Comparing The Performance Of Two Different Daily Disposable Lenses (MIKI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-114
Record Dates: First submitted 2020-07-24; First posted 2020-07-30 (Actual); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test Contact lens (Experimental): Subjects will be randomized to wear test lenses for one week and then switch to control lenses for one week.
  Interventions: Device: Test Contact Lens; Device: Control Contact Lens
- Control Contact Lens (Active Comparator): Subjects will be randomized to wear control lenses for one week and then switch to test lenses for one week.
  Interventions: Device: Test Contact Lens; Device: Control Contact Lens

INTERVENTIONS:
Device: Test Contact Lens — Subjects will be randomized to wear test lenses.
  Other Names: stenfilcon A
Device: Control Contact Lens — Subjects will be randomized to wear control lenses.
  Other Names: verofilcon A

SUMMARY:
The objective of the study is to evaluate and compare the performance of study test lens to study control lens, when worn on a daily disposable modality over a period of approximately one week each

DETAILED DESCRIPTION:
The study is a prospective, double masked (investigator and participant), bilateral, randomized,one week cross-over dispensing study, which evaluates the study test lens and control lens.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 17 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Habitually wears soft contact lenses in daily wear, for minimum of 6-months;
5. Is correctable to a visual acuity of 20/40 or better (in each eye) with the study lenses;
6. Has an astigmatism of ≤ 1.00 D in subjective refraction;
7. Can be fit with study contact lenses with a power between -2.00 and -5.00 DS;
8. Demonstrates an acceptable fit with the study lenses;
9. Habitually wears single vision soft contact lenses for at least 8 hours per day, 5 days a week, and is willing to wear contact lenses for at least 12 hours a day in the study.

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Has any known active* ocular disease and/or infection;
3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
5. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
6. Is pregnant, lactating or planning a pregnancy at the time of enrolment because the associated hormonal changes cause changes in the tear layer which impact contact lens comfort. Verbal confirmation at the screening visit is sufficient;
7. Is aphakic;
8. Has undergone refractive error surgery;
9. Is an employee of the Centre for Ocular Research & Education;
10. Has participated in the BOXER (i.e. EX-MKTG-107, phases 1 or 2) or BASSET (EXMKTG-113) Study;
11. Has participated in any clinical trials within a week prior to the study.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD FCOptom, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty-one subjects were screened and 35 subjects started and completed the study.
Groups:
- Test Contact Lens the Control Contact Lens: Subjects will be randomized to wear test lenses for one week and then switch to control lenses for one week.
  Test Contact Lens: Subjects will be randomized to wear test lenses.
  Control Contact Lens: Subjects will be randomized to wear control lenses.
- Control Contact Lens Then Test Contact Lens: Subjects will be randomized to wear control lenses for one week and then switch to test lenses for one week.
  Test Contact Lens: Subjects will be randomized to wear test lenses.
  Control Contact Lens: Subjects will be randomized to wear control lenses.
Period: First Intervention
Arm/Group | Test Contact Lens the Control Contact Lens | Control Contact Lens Then Test Contact Lens
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Test Contact Lens the Control Contact Lens | Control Contact Lens Then Test Contact Lens
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Forty-one subjects were screened and demographic data includes all screened subjects.
Groups:
- Overall Study: Subjects will be randomized to wear control lenses and test lenses for one week.
  Contact lenses: Test Contact Lens Contact lenses: Control Contact Lens
Arm/Group | Overall Study
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 39
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 41

OUTCOME MEASURES:

1. Primary Outcome: Overall Lens Fit Acceptance
Description: Overall fit acceptance (0-4, 0.50 steps) (0 - lens should not be worn at all,1 - Borderline but unacceptable, 2 - Minimally acceptable, 3 - Not perfect but OK to dispense, 4 - Perfect)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Test Contact Lens: Subjects will be randomized to wear test lenses for one week and then switch to control lenses for one week.
  Contact lenses: Test Contact Lens
- Control Contact Lens: Subjects will be randomized to wear control lenses for one week and then switch to test lenses for one week.
  Contact lenses: Control Contact Lens
Arm/Group | Test Contact Lens | Control Contact Lens
Number analyzed (Participants) | 35 | 35
units on a scale | 3.71 (0.33) | 3.73 (0.35)

2. Secondary Outcome: Lens Centration
Description: Lens Centration was measured on a scale (0-3) (0 = "Optimally centered", 1 = "Slightly decentered", 2 = Moderate decentration but not encroaching limbus, 3 = "Excessive & occasionally encroaching limbus")
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Contact Lens | Control Contact Lens
Number analyzed (Participants) | 35 | 35
units on a scale | 0.40 (0.50) | 0.29 (0.52)

3. Secondary Outcome: Lens Centration
Description: as for outcome 2
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Contact Lens | Control Contact Lens
Number analyzed (Participants) | 35 | 35
units on a scale | 0.17 (0.38) | 0.20 (0.47)

4. Secondary Outcome: Post-blink Movement
Description: Post-blink lens movement was measured using an eyepiece reticule while viewing the contact lens in-vivo at 8x magnification in primary gaze, in 0.1mm steps
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Test Contact Lens | Control Contact Lens
Number analyzed (Participants) | 35 | 35
mm | 0.20 (0.06) | 0.23 (0.06)

5. Secondary Outcome: Post-blink Movement
Description: as for outcome 4
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Test Contact Lens | Control Contact Lens
Number analyzed (Participants) | 35 | 35
mm | 0.20 (0.05) | 0.23 (0.07)

6. Secondary Outcome: Push-up Tightness
Description: Push-up tightness in primary gaze measured on a scale (0-100, 5% steps) (0% = falls from cornea without lid support, 50% = optimum, 100% = no movement)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Contact Lens | Control Contact Lens
Number analyzed (Participants) | 35 | 35
units on a scale | 51 (5) | 49 (6)

7. Secondary Outcome: Push-up Tightness
Description: Push-up tightness in primary gaze measured on a scale (0-100, 5% steps) (0% = falls from cornea without lid support, 50% = optimum and 100% = no movement)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Contact Lens | Control Contact Lens
Number analyzed (Participants) | 35 | 35
units on a scale | 50 (4) | 48 (4)

ADVERSE EVENTS:
Time Frame: From dispense up to 1 week for a total of 2 weeks
Arm/Group | Test Contact Lens | Control Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT04492397/Prot_SAP_000.pdf